CLINICAL TRIAL: NCT05327166
Title: The Emergency Department Longitudinal Integrated Care Effectiveness Randomized Trial Targeting Opioid Use and Related Comorbidity From the ED
Brief Title: The Emergency Department Longitudinal Integrated Care
Acronym: ED-LINC2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren Whiteside, Assistant Professor, Department of Emergency Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00012599; R01DA051462 (NIH)
Record Dates: First submitted 2022-02-18; First posted 2022-04-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
Keywords: collaborative care; opioid use disorder (OUD); substance use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either usual care (n=250) or ED-LINC intervention (n=250). Patients assigned to the ED-LINC intervention will receive 1) overdose education, 2) brief bedside intervention targeting motivation to engage in outpatient care, 3) a patient-centered approach to MOUD using a treatment decision support tool, 4) longitudinal and proactive care management which will proceed for 3 months, and 5) weekly caseload supervision allowing for stepped-up care targeting opioid use and comorbidity.
Masking Description: Due to the nature of the intervention, this is an open label study since participants will know whether they are receiving ED-LINC resources or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants assigned to this arm will receive usual care.
- ED-LINC Intervention (Experimental): Patients assigned to the ED-LINC intervention will receive 1) overdose education, 2) brief bedside intervention targeting motivation to engage in outpatient care, 3) a patient-centered approach to MOUD using a treatment decision support tool, 4) longitudinal and proactive care management and 5) weekly caseload supervision allowing for stepped-up care targeting opioid use and comorbidity.
  Interventions: Other: ED-LINC

INTERVENTIONS:
Other: ED-LINC — The ED-LINC intervention provides 1) overdose education, 2) brief bedside intervention targeting motivation to engage in outpatient care, 3) a patient-centered approach to MOUD using a treatment decision support tool, 4) longitudinal and proactive care management which will proceed for 3 months, and 5) weekly caseload supervision allowing for stepped-up care targeting opioid use and comorbidity.
  Other Names: Collaborative Care
  Arms: ED-LINC Intervention

SUMMARY:
Collaborative care is a comprehensive patient-centered model of healthcare delivery targeting behavioral health or substance use that stems from the chronic disease management framework. The intervention being tested ('Emergency Department Longitudinal Integrated Care' or ED LINC) derives from the collaborative care model and has demonstrated feasibility in previous studies.

This study expands on the model to test the effectiveness of the ED-LINC intervention when compared with usual care. The study team primarily hypothesizes that patients randomized to the ED-LINC intervention, when compared to patients randomized to usual care, will demonstrate: 1) significant reductions in self-report illicit opioid use, 2) significant increases in initiation and retention of medications for opioid use disorder, and 3) significant reductions in ED utilization.

DETAILED DESCRIPTION:
This is a randomized clinical trial designed to test the effectiveness of the multi-component ED-LINC intervention. Patients with moderate or severe OUD seeking medical care at 2 EDs in Seattle, Washington, who provide informed consent will be randomized to the ED-LINC intervention (n=250) or usual care control (n=250) conditions.

ED-LINC will include: 1) overdose education, 2) brief bedside intervention targeting motivation to engage in outpatient care, 3) a patient-centered approach to medications for opioid use disorder (MOUD) using a treatment decision support tool, 4) longitudinal and proactive care management which will proceed for approximately 3 months, and 5) weekly caseload supervision allowing for stepped-up care targeting opioid use and comorbidity. This intervention will use the Emergency Department Information Exchange (EDIE) to re-engage patients with subsequent ED visits.

This study team developed the 'Emergency Department Longitudinal Integrated Care 2.0' intervention or 'ED-LINC' for patients with OUD to be initiated from the ED. In prior work, ED-LINC was feasible and retention in the study was high in both an intervention arm and a usual care control arm. Additionally, participants randomized to the ED-LINC arm were satisfied and acceptability of the intervention was high. Elements of ED-LINC are based on evidence-based treatments and are central components of collaborative care and will acknowledge the longitudinal care required for opioid use disorder and related substance abuse, mental health and medical comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Moderate or Severe OUD based on the Structured Clinical Interview for DSM Disorders (SCID)
* Currently have a phone or method of contact
* Able to provide a phone number and one additional piece of contact information

Exclusion Criteria:

* Incarcerated or under arrest
* Non-English speaking
* Live beyond a 50 mile radius of Harborview Medical Center
* Require active resuscitation in the ED or other clinical area at the time of Research Assistant (RA) approach
* Are receiving palliative care services or hospice care for a chronic illness such as metastatic cancer
* Are in the ED or hospital for a primary psychiatric emergency such as suicidal ideation or attempt and require emergent evaluation by a Psychiatrist
* Receiving chronic opioid therapy (COT) defined as prescription opioids for most days out of the last 90 days for a chronic pain condition
* In the ED for sexual assault
* Enrolled or eligible for state-funded or hospital-funded care coordination program based on high utilization of the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Illicit Opioid Use Over Time | Baseline ED visit and 1, 3, 6 and 12-months after ED visit
  To compare self-reported past-30 day illicit opioid use using the validated self-report measure of timeline followback (TLFB) in subjects receiving usual care or ED-LINC intervention over the course of the year after the index Emergency Department visit.
Initiation of Medications for OUD | 12 months
  To compare the frequency of initiation of medications for opioid use disorder (MOUD) where MOUD includes buprenorphine, methadone and/or naltexone in subjects receiving usual care or ED-LINC intervention over the course of the year after the index Emergency Department visit using statewide data for prescriptions and Medicaid billing data for medication administration augmented with patient self-report MOUD at scheduled follow-up intervals.
Change in Emergency Department visits | Index Emergency Department visit to 12-months followup
  To compare changes over time in Emergency Department visits in subjects receiving usual care or ED-LINC intervention; Emergency Department visits will be measured by the Emergency Department Information Exchange (an automated health information exchange) that caputures population-level Emergency Department utilization for all enrolled participants.

SECONDARY OUTCOMES:
Intervention effect when associated with Methamphetamine use | Index Emergency Department visit to 12-months followup
  Explore the impact of methamphetamine use, as measured by the timeline follow-back (TLFB) which is a validated patient self-report measure of days of methamphetamine use over a 30 day-period, on intervention treatment effects.
Time to Initiation of MOUD | 12 months
  To compare time to initiation of medications for opioid use disorder (MOUD) where MOUD includes buprenorphine, methadone and/or naltexone in subjects receiving usual care or ED-LINC intervention over the course of the year after the index Emergency Department visit.
Engagement in Medications for OUD | 12 months
  To compare the frequency of engagement in medications for opioid use disorder (MOUD) where MOUD includes buprenorphine, methadone and/or naltexone in subjects receiving usual care or ED-LINC over the course of the year after the index Emergency Department visit using statewide data for prescriptions and Medicaid billing data for medication administration augmented with patient self-report MOUD at scheduled follow-up intervals.
Retention in Medications for OUD | 12 months
  To compare the frequency of retention in medications for opioid use disorder (MOUD) where MOUD includes buprenorphine, methadone and/or naltexone in subjects receiving usual care or ED-LINC intervention over the course of the year after the index Emergency Department visit visit using statewide data for prescriptions and Medicaid billing data for medication administration augmented with patient self-report MOUD at scheduled follow-up intervals.
Intervention effect when associated depression | Index Emergency Department visit to 12-months followup
  Explore the impact of depression in the past 30-days as measured by self-report PHQ-9 at baseline on intervention treatment effects.
Intervention effect when associated anxiety | Index Emergency Department visit to 12-months followup
  Explore the impact of anxiety in the past 30-days as measured by self-report GAD-7 at baseline on intervention treatment effects.
Intervention effect when associated PTSD | Index Emergency Department visit to 12-months followup
  Explore the impact of PTSD in the past 30-days as measured by self-report PCL-C at baseline on intervention treatment effects.baseline on intervention treatment effects.
Intervention effect when associated current pain | Index Emergency Department visit to 12-months followup
  Explore the impact of pain in the past week as measured by the self-report 3-item PEG at baseline on intervention treatment effects.
Intervention effect when patient has exposure to MOUD in prior 12 months | Index Emergency Department visit to 12-months followup
  Explore the impact of any past 12-month MOUD exposure prior to enrollment where MOUD includes buprenorphine, methadone and/or naltexone assessed from review of medical records, using statewide data for prescriptions and Medicaid billing data for medication administration augmented with patient self-report MOUD obtained at baseline on the intervention treatment effect.
Intervention effect by sex | Index Emergency Department visit to 12-months followup
  Explore the impact of patient sex as measured by patient self-report at baseline on intervention treatment effects
Intervention effect when patient reports using illicit fentanyl at baseline | Index Emergency Department visit to 12-months followup
  Explore the impact of fentanyl use as measured by any patient self-report fentanyl use in the past 30-days at baseline on the intervention treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Lauren K Whiteside, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States